CLINICAL TRIAL: NCT06399497
Title: Effects of Lumbar Spinal Manipulation on Muscle Mechanical Properties, Pressure Pain Threshold and Mechanical Perception Threshold in Subjects With Chronic Low Back Pain
Brief Title: Effects of Lumbar Spinal Manipulation in Subjects With Chronic Low Back Pain
Acronym: LBP-HVLA
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Córdoba (Other)
Responsible Party: Principal Investigator, Lourdes García Luque, Principal Investigator, Universidad de Córdoba
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 5874
Record Dates: First submitted 2024-04-30; First posted 2024-05-03 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Low Back Pain
Keywords: Manipulation, Spinal; Muscle Mechanical Properties; Pain Threshold; Perception Threshold
MeSH Terms: conditions — Low Back Pain | interventions — Manipulation, Spinal; Heimlich Maneuver

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The assessor will be blinded to the intervention assigned to each participant.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group (Experimental): A physical therapist, with more than 10 years of experience, performs a high-velocity low-amplitude spinal manipulation at the L5 level by means of the lumbar roll technique, performed with the subject in right lateral decubitus.
  Interventions: Other: spinal manipulation
- Control Group (Placebo Comparator): A physical therapist performance a simulated manipulation intervention, for which the same position as in the Intervention Group will be used, in right lateral decubitus with the left leg flexed and the left foot resting on the right popliteal fossa. Without stretching the paravertebral tissues, the participant will remain for approximately 20 seconds without receiving manual impulse.
  Interventions: Other: simulated manipulation

INTERVENTIONS:
Other: spinal manipulation — A high-velocity low-amplitude spinal manipulation at the L5 level will be performance by means of the lumbar roll technique, with the subject in right lateral decubitus.
  Other Names: thrust; high-velocity low-amplitude
  Arms: Intervention Group
Other: simulated manipulation — Simulated manipulation intervention, in the same position as in the Intervention Group, performance in right lateral decubitus with the left leg flexed and the left foot resting on the right popliteal fossa. Without stretching the paravertebral tissues, the participant will remain for approximately 20 seconds without receiving manual impulse.
  Other Names: placebo intervention
  Arms: Control Group

SUMMARY:
This study aims to measure the effects of spinal manipulation on Chronic Spinal Pain by assessing Muscle Mechanical Properties (MMPs) using MyotonPRO®, Mechanical Perception Threshold (MPT) using Von Frey monofilaments, and Pressure Pain Threshold (PPT) using an algometer. Participants will be randomly assigned to either spinal manipulation or placebo groups to compare effects on MMPs, MPT, and PPT. Assessments will occur at three time points: baseline, immediately post-intervention (real or simulated), and 24 hours post-intervention. This research targets individuals with chronic spinal pain, providing insights into the potential benefits of spinal manipulation in managing this condition.

ELIGIBILITY:
Inclusion Criteria:

* Subject with chronic low back pain

Exclusion Criteria:

* Spinal trauma or surgery history.
* Spinal congenital deformities.
* Inflammatory or autoimmune disease
* Herniated disc in the segment L5.
* Pregnant women.
* Body Mass Index > 30kg/m2
* Subjects that have received treatment for low back pain in the seven days prior to the study.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Estimated)
Dates: Start 2024-05 (Estimated); Primary Completion 2025-05 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Muscle mechanical propierties | From enrollment to the end of treatment at 24 hours
  The measurements will be performed with the MyotonPro®. The subject will be positioned in prone position with both upper limbs around the body. They will be asked to breathe apnea for five seconds after exhaling to reduce the abdominal influence on the test. Measurements at the lumbar level will be performed by positioning the MyotonPro® probe perpendicular to the muscle belly of the erector spinae, 2.5 cm from the midline of the spinous process of L5. A measurement of the tibialis anterior will assess the effect of the remote manipulation. For this purpose, the subject will be positioned in supine decubitus with the lower limb in extension. A point will be located on the tibialis anterior muscle, three finger traverses from the crest of the tibia in a caudal direction.

SECONDARY OUTCOMES:
Pressure pain threshold | From enrollment to the end of treatment at 24 hours
  An Algometer Commander™ JTECH will be used. Prior to the measurements, the subject will be familiarized with the evaluation by taking three measurements in the tenar region of the hand. During this phase, the subject will be asked to indicate, with eyes closed, the moment in which he perceives the painful sensation. The test will consist of a combination of three measurements administered to each muscle, with an interval between measurements of 3 to 5 seconds. The pressure stimulation will be applied with an algometer, gradually increasing the pressure by 0.5 kg per second until the subject manifests pain. The mean pressure at which the subject manifested pain will be calculated from these three measurements. The algometer will be placed perpendicular to the muscle bellies, and the subject will maintain the same position as in the measurement of the muscle mechanical propierties. The evaluation locations will be the L5 spinal Level and the tibialis anterior (bilaterally)
Mechanical perception threshold | From enrollment to the end of treatment at 24 hours
  It will be evaluated by means of Von Frey monofilaments, which will be applied perpendicularly to the cutaneous surface, with ascending diameter consecutively until the patient reports tactile perception. Prior to the measurements, the subject will be familiarized with the evaluation by taking three measurements in the tenar region of the hand. During this phase, the subject will be asked to indicate, with eyes closed, the moment in which he perceives the pressure sensation. The evaluation sites will be the same as in the MMPs: L5 level. Anterior tibial (bilaterally).

CONTACTS AND LOCATIONS:
Overall Officials: Lourdes García Luque, PhD, Principal Investigator — Universidad de Córdoba
Locations (1):
- Physiobalance, Córdoba, Spain

IPD SHARING:
Plan to Share IPD: Undecided
The investigators have decided to first present the data in different forums and journals before making the database available

REFERENCES:
- [Background] Trierweiler J, Gottert DN, Gehlen G. Evaluation of mechanical allodynia in an animal immobilization model using the von frey method. J Manipulative Physiol Ther. 2012 Jan;35(1):18-25. doi: 10.1016/j.jmpt.2011.09.007. Epub 2011 Nov 4. PMID 22054875
- [Background] Tracey EH, Greene AJ, Doty RL. Optimizing reliability and sensitivity of Semmes-Weinstein monofilaments for establishing point tactile thresholds. Physiol Behav. 2012 Feb 28;105(4):982-6. doi: 10.1016/j.physbeh.2011.11.002. Epub 2011 Nov 11. PMID 22100625
- [Background] Keizer D, van Wijhe M, Post WJ, Wierda JM. Quantifying allodynia in patients suffering from unilateral neuropathic pain using von frey monofilaments. Clin J Pain. 2007 Jan;23(1):85-90. doi: 10.1097/01.ajp.0000210950.01503.72. PMID 17277649
- [Background] Garcia-Perez-Juana D, Fernandez-de-Las-Penas C, Arias-Buria JL, Cleland JA, Plaza-Manzano G, Ortega-Santiago R. Changes in Cervicocephalic Kinesthetic Sensibility, Widespread Pressure Pain Sensitivity, and Neck Pain After Cervical Thrust Manipulation in Patients With Chronic Mechanical Neck Pain: A Randomized Clinical Trial. J Manipulative Physiol Ther. 2018 Sep;41(7):551-560. doi: 10.1016/j.jmpt.2018.02.004. PMID 30442354
- [Background] Nogueira N, Oliveira-Campelo N, Lopes A, Torres R, Sousa ASP, Ribeiro F. The Acute Effects of Manual and Instrument-Assisted Cervical Spine Manipulation on Pressure Pain Threshold, Pressure Pain Perception, and Muscle-Related Variables in Asymptomatic Subjects: A Randomized Controlled Trial. J Manipulative Physiol Ther. 2020 Mar-Apr;43(3):179-188. doi: 10.1016/j.jmpt.2019.05.007. PMID 32951766
- [Background] Lohr C, Braumann KM, Reer R, Schroeder J, Schmidt T. Reliability of tensiomyography and myotonometry in detecting mechanical and contractile characteristics of the lumbar erector spinae in healthy volunteers. Eur J Appl Physiol. 2018 Jul;118(7):1349-1359. doi: 10.1007/s00421-018-3867-2. Epub 2018 Apr 20. PMID 29679246
- [Background] Dellalana LE, Chen F, Vain A, Gandelman JS, Poldemaa M, Chen H, Tkaczyk ER. Reproducibility of the durometer and myoton devices for skin stiffness measurement in healthy subjects. Skin Res Technol. 2019 May;25(3):289-293. doi: 10.1111/srt.12646. Epub 2018 Nov 10. PMID 30414198
- [Background] Kurashina W, Iijima Y, Sasanuma H, Saito T, Takeshita K. Evaluation of muscle stiffness in adhesive capsulitis with Myoton PRO. JSES Int. 2022 Sep 17;7(1):25-29. doi: 10.1016/j.jseint.2022.08.017. eCollection 2023 Jan. PMID 36820433
- [Background] Wu Z, Zhu Y, Xu W, Liang J, Guan Y, Xu X. Analysis of Biomechanical Properties of the Lumbar Extensor Myofascia in Elderly Patients with Chronic Low Back Pain and That in Healthy People. Biomed Res Int. 2020 Feb 18;2020:7649157. doi: 10.1155/2020/7649157. eCollection 2020. PMID 32149135
- [Background] Ilahi S, T Masi A, White A, Devos A, Henderson J, Nair K. Quantified biomechanical properties of lower lumbar myofascia in younger adults with chronic idiopathic low back pain and matched healthy controls. Clin Biomech (Bristol). 2020 Mar;73:78-85. doi: 10.1016/j.clinbiomech.2019.12.026. Epub 2020 Jan 2. PMID 31954272
- [Background] Dorron SL, Losco BE, Drummond PD, Walker BF. Effect of lumbar spinal manipulation on local and remote pressure pain threshold and pinprick sensitivity in asymptomatic individuals: a randomised trial. Chiropr Man Therap. 2016 Dec 5;24:47. doi: 10.1186/s12998-016-0128-5. eCollection 2016. PMID 27980726
- [Background] Jun P, Page I, Vette A, Kawchuk G. Potential mechanisms for lumbar spinal stiffness change following spinal manipulative therapy: a scoping review. Chiropr Man Therap. 2020 Mar 23;28(1):15. doi: 10.1186/s12998-020-00304-x. PMID 32293493
- [Background] Page I, Descarreaux M. Effects of spinal manipulative therapy biomechanical parameters on clinical and biomechanical outcomes of participants with chronic thoracic pain: a randomized controlled experimental trial. BMC Musculoskelet Disord. 2019 Jan 18;20(1):29. doi: 10.1186/s12891-019-2408-4. PMID 30658622
- [Background] Fagundes Loss J, de Souza da Silva L, Ferreira Miranda I, Groisman S, Santiago Wagner Neto E, Souza C, Tarrago Candotti C. Immediate effects of a lumbar spine manipulation on pain sensitivity and postural control in individuals with nonspecific low back pain: a randomized controlled trial. Chiropr Man Therap. 2020 Jun 3;28(1):25. doi: 10.1186/s12998-020-00316-7. PMID 32487243